CLINICAL TRIAL: NCT03893045
Title: A Phase 3, Randomized, Open-Label, Multicenter Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Ferumoxytol for the Treatment of Iron Deficiency Anemia (IDA) in Pediatric Subjects
Brief Title: A Study to Evaluate Ferumoxytol for the Treatment of Iron Deficiency Anemia (IDA) in Pediatric Subjects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-IDA-352
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Iron Deficiency Anemia
Keywords: IDA; anemia; pediatrics; ferumoxytol; iron sucrose
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — Ferrosoferric Oxide; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferumoxytol (Experimental): Each 20 mL single-use vial contains 17 mL of ferumoxytol that consists of iron at a concentration of 30 mg Fe/mL, coated with polyglucose sorbitol carboxymethylether and formulated with mannitol, at a concentration of 44 mg/mL, in a black to reddish brown sterile, aqueous, colloidal, isotonic solution.
  Interventions: Drug: ferumoxytol
- Iron sucrose (Active Comparator): Each mL contains 20 mg of elemental iron as iron sucrose in water for injection. The 5 mL single-use vial contains 100 mg of iron per 5 mL. The drug product contains approximately 30% sucrose (300 mg/mL)
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: ferumoxytol — Each 20 mL single-use vial contains 17 mL of ferumoxytol that consists of iron at a concentration of 30 mg Fe/mL, coated with polyglucose sorbitol carboxymethylether and formulated with mannitol, at a concentration of 44 mg/mL, in a black to reddish brown sterile, aqueous, colloidal, isotonic solution
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: Iron sucrose — Each mL contains 20 mg of elemental iron as iron sucrose in water for injection. The 5 mL single-use vial contains 100 mg of iron per 5 mL. The drug product contains approximately 30% sucrose (300 mg/mL).
  Other Names: Venofer
  Arms: Iron sucrose

SUMMARY:
This is a Phase 3, randomized, open-label, multicenter, study in male and female pediatric subjects (2 years to <18 years of age) with IDA, or felt by their clinician to be at risk of developing IDA. This study allows for enrollment of subjects with IDA regardless of etiology, except for CKD subjects (pediatric CKD subjects are being studied in a separate ferumoxytol protocol).

DETAILED DESCRIPTION:
Subjects will be randomized to treatment in a 2:1 ratio (ferumoxytol: iron sucrose) and stratified by age group (2 to <6 years; 6 to <12 years; and 12 to <18 years). Subjects will receive one of the following treatment regimens:

• Ferumoxytol: 7 mg Fe/kg IV (maximum 510 mg/dose) x 2 doses, the first dose administered on Day 1 and the second 2 to 8 days later.

OR

• Iron sucrose (Venofer®): 4 mg Fe/kg IV (maximum 200 mg/dose) x 5 doses, the first dose on Day 1 and subsequent doses administered at least once per week and up to 3 times/week. All subjects will be monitored at the study site through at least 1 hour after the completion of each infusion of study drug. Assessment of blood Hgb concentrations, adverse events, and other safety assessments will be performed through study Week 5.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 2 years to <18 years of age at time of consent
2. Has IDA defined as:

   1. Hemoglobin (Hgb) <11.0 g/dL AND
   2. Any one or more of the following:

      * Transferrin saturation (TSAT) <20%
      * ferritin <100 ng/mL
3. Documented history of unsatisfactory oral iron therapy or in whom oral iron cannot be tolerated, or for whom oral iron is considered medically inappropriate

Exclusion Criteria:

1. Known hypersensitivity reaction to any component of ferumoxytol or iron sucrose
2. History of allergy to intravenous (IV) iron
3. History of ≥2 clinically significant drug allergies
4. Subjects with CKD (defined as eGFR of <60 mL/min/1.73 m2 or a requirement for chronic hemodialysis or peritoneal dialysis during Screening)
5. Low systolic blood pressure (BP) (age 1 to 9 years <70 + [age in years x 2] mmHg, age 10 to 17 years <90 mmHg)
6. Hgb ≤7.0 g/dL
7. Serum ferritin level >600 ng/mL

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin from Baseline to Week 5 | 35 days
  Proportion of subjects achieving a change in hemoglobin from Baseline to Week 5

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 49 days
  Incidence of Treatment Emergent Adverse Events
Incidence of adverse events of special interest (AESI) | 49 days
  Incidence of adverse events of special interest (AESI) (hypotension and hypersensitivity)

OTHER OUTCOMES:
Area Under the Curve (AUC) | 35 days
  Pharmacokinetic parameter: Area Under the Curve (AUC)
Clearance | 35 days
  Pharmacokinetic parameter: Clearance
Distribution | 35 days
  Pharmacokinetic parameter: Distribution
Elimination half-lives | 35 days
  Pharmacokinetic parameter: Elimination half-lives

CONTACTS AND LOCATIONS:
Locations (15):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida
  - Optimus U Corporation, Miami, Florida
  - Biomedical Research LLC, Miami, Florida
  - Gwinnett Research Institute, Buford, Georgia
  - Sun Research Institute, San Antonio, Texas
- Lithuania (3):
  - JSC Saules seimos medicinos centras, Kaunas
  - Klaipeda Children's Hospital, Klaipėda
  - Children's Hospital-Affiliate of Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Poland (6):
  - Osrodek Badan Klinicznych In Vivo sp. z o.o., Bydgoszcz
  - Prywatny Gabinet Lekarski Dr N. med. Jerzy Brzostek, Dębica
  - Pro Familia Altera Sp. z o.o., Katowice
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Centrum Zdrowia MDM, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: No